

# TRIAL STATISTICAL ANALYSIS PLAN

c10164918-03

BI Trial No.: 1315.2

Title: An open-label, Phase I/II trial to determine the maximum tolerated

dose and investigate safety, pharmacokinetics and efficacy of BI 836858 in combination with decitabine in patients with acute

myeloid leukemia

Including:

Protocol Amendment 1 [c03377067-02] Protocol Amendment 2 [c03377067-03] Protocol Amendment 3 [c03377067-04] Protocol Amendment 4 [c03377067-05] Protocol Amendment 5 [c03377067-06] Protocol Amendment 6 [c03377067-07]

Investigational Product(s):

BI 836858

Responsible trial statistician(s):



Fax:

Date of statistical analysis plan:

19NOV 2019 SIGNED

\_\_\_\_\_

Version: Final

Page 1 of 33

**Proprietary confidential information** 

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

| 4 | ADI | | OE | 00 | TIT | 1 | TOO |
|----|-----|------|----|----|-----|-----|-----|
| I. | ABI | , H, | OF | CU | | H.I | 115 |

| | TIBLE OF CONTENTS |
|-------------|--------------------------------------------------|
| TITLE PAGE1 | |
| 1. | TABLE OF CONTENTS2 |
| LIST OF | ΓABLES4 |
| 2. | LIST OF ABBREVIATIONS5 |
| 3. | INTRODUCTION8 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY9 |
| 5. | ENDPOINTS(S)9 |
| 5.1 | PRIMARY ENDPOINT(S)9 |
| 5.2 | SECONDARY ENDPOINT(S)9 |
| 5.2.1 | Key secondary endpoint(s)9 |
| 5.2.2 | Secondary endpoint(s)9 |
| 6. | GENERAL ANALYSIS DEFINITIONS12 |
| 6.1 | TREATMENT(S) |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS |
| 6.3 | SUBJECT SETS ANALYSED |
| 0.0 | |
| 6.5 | POOLING OF CENTRES16 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS16 |
| 6.7 | BASELINE, TIME WINDOWS AND CALCULATED VISITS16 |
| 7. | PLANNED ANALYSIS |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS18 |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION19 |
| 7.3 | TREATMENT COMPLIANCE |
| 7.4 | PRIMARY ENDPOINT(S) |
| 7.5 | SECONDARY ENDPOINT(S) |
| 7.7 | EXTENT OF EXPOSURE20 |
| 7.8 | SAFETY ANALYSIS |
| 7.8.1 | Adverse Events20 |
| 7.8.2 | Laboratory data |
| 7.8.3 | Vital signs |
| 7.8.4 | ECG |

| 8. | REFERENCES | 31 |
|----|---------------|----|
| 10 | HISTORY TARLE | 33 |

# LIST OF TABLES

| Table 6.1:1 | Definition of analysing treatment periods | 13 |
|---|---|---|
| Table 6.2:1 | Important protocol deviations | 14 |
| Table 7.8.1:1 | Definition of user-defined AE categories | 22 |
| | User-defined (sub-) search category of "Cardiac Failure" | |
| Table 7.8.1:3 | Laboratory Signs of Cell Destruction | 26 |
| | Clinical Signs of Cell Destruction | |
| | History table | |

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|--------------------|------------------------------------------------------|
| AE | Adverse event |
| AESI | Adverse events of special interest |
| ALKP | Alkaline phosphatase |
| ALT | Alkaline aminotransferase |
| AST | Aspartate aminotransferase |
| ATC classification | Anatomical, Therapeutic, Chemical classification |
| AUC | Area Under Curve |
| BI | Boehringer Ingelheim |
| BLRM | Bayesian logistic regression model |
| BSA | Body Surface Area |
| RPM | Report planning meeting |
| $C_{max}$ | Maximum measured plasma concentration of the analyte |
| CL | Total plasma clearance |
| CR | Complete Remission |
| CRi | Complete Remission with incomplete marrow recovery |
| CT | Concomitant therapy |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| DBL | Data Base Lock |
| DILI | Drug Induced Liver Injury |
| DLT | Dose Limiting Toxicity |
| DMS | Data Management and Statistics |
| DOR | Duration of Remission |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eDISH | Evaluation of Drug Induced Serious Hepatotoxicity |
| EFS | Event free survival |
| eCRF | Electronic case report form |
| ICH | International Conference on Harmonisation |

| Term | Definition / description |
|---|---|
| iPD | Important Protocol Deviation |
| IRR | Infusion Related Reaction |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MQRM | Medical and Quality Review Meeting |
| MTD | Maximum tolerated dose |
| NE | Not evaluable |
| OR | Objective response |
| OS | Overall survival |
| PD | Progressive disease |
| PFS | Progression free survival |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic set |
| PR | Partial remission |
| PT | Preferred term |
| PV | Protocol deviation |
| REP | Residual effect period |
| REPd | Duration of residual effect period in days |
| RFS | Relapse free survival |
| RP2D | Recommended phase 2 dose |
| RPM | Report planning meeting |
| SAE | Serious adverse event |
| SD | Standard deviation |
| SOC | System organ class |
| SOP | Standard Operating Procedure |
| SS | Screened set |
| TCM | Trial Clinical Monitor |
| TF | Treatment failure |
| $t_{max}$ | Time from dosing to the maximum plasma concentration of the analyte |
| TOC | Table of contents |
| TS | Treated set |

| Term | Definition / description |
|------|---------------------------|
| TTF | Time to treatment failure |

# 3. INTRODUCTION

As per ICH E9(1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the protocol, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the Clinical Trial Protocol (CTP), including Protocol Amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation. This TSAP follows the Boehringer Ingelheim (BI) internal reference (2).

This TSAP is based on the Project SAP wherever possible. Wordings like "randomisation (first administration of study treatment in non-randomised trials)" should therefore be interpreted as applicable.

Furthermore, in this combination trial the term investigational medicinal product is used for BI 836858 while combination drug denotes the backbone chemotherapy decitabine. The term trial medication is used for any of the two trial drugs.

SAS Version 9.4 or later version will be used for all analyses.

Due to company decision to stop this project, there is no Phase II subject enrollment so that Phase II analyses stated in CTP will be omitted.

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

Due to the decision to discontinue the development of BI865868, the enrollment was stopped after Phase I extension and Phase II part of the trial was cancelled as stated in CTP amendment 7.0. Thus there will be no data collection nor analyses for Phase II part .

# 5. ENDPOINTS(S)

# 5.1 PRIMARY ENDPOINT(S)

#### Phase I

The primary endpoints in the Phase I part of the trial are the maximum tolerated dose (MTD) and the number of subjects with of dose limiting toxicity (DLT) during the MTD evaluation period.

## Maximum tolerated dose (MTD):

The MTD is defined as the highest dose of BI 836858 (in combination with decitabine) with less than 25% risk of the true DLT rate being above 33% during the MTD evaluation period.

# MTD evaluation period:

The MTD evaluation period is defined as the time from the first administration of study drug to the start of the second treatment cycle or the end of 30-day residual effect period after last administration of study drug, whichever comes first. Subjects who were replaced during the MTD evaluation period will not be considered for MTD determination. The subjects who are completed the MTD evaluation period without being replaced are considered MTD evaluable.

In case a subject has not completed the required number of administrations due to BI 836858 related toxicity, he/she will not be replaced and this will be considered as DLT. However, subjects who have not completed the required number of administrations of BI 836858 for reasons other than BI 836858 related toxicity will be replaced. Subjects who were replaced during the MTD evaluation period will not be considered for MTD

# 5.2 SECONDARY ENDPOINT(S)

# 5.2.1 Key secondary endpoint(s)

No key secondary endpoints are defined in this study.

### 5.2.2 Secondary endpoint(s)

# Phase I

- Number of subjects with objective response combining
  - Complete remission (CR)
  - CR with incomplete blood count recovery (CRi)

• Time frame: From start of treatment until the earliest of progression, death or end of trial (approximately up to 30 months).







- **GENERAL ANALYSIS DEFINITIONS 6.**
- 6.1 **TREATMENT(S)**

Phase I

In the Phase I Part, treatments are not randomized (open-label, dose escalation). Different dose levels of the investigational medicinal product (BI 836858) can arise while combined with fixed dose of decitabine at 20 mg/m² per day. The data will be presented for all dose cohorts separately, in particular, subjects will be analysed by the dose cohort initially assigned in the first treatment course.

Table 6.1:1 Definition of analysing treatment periods

| Analysing treatment period | Start date (including) | Stop date (excluding) |
|---|---|---|
| Screening | Date of informed consent | Date of first administration of trial medication |
| MTD evaluation period | Date of first<br>administration of trial<br>medication | First of start of the second treatment cycle or the end of the 30-day residual effect period |
| On-treatment | Date of first<br>administration of trial<br>medication | Start date of 'Follow-up' |
| Follow-up | Date of end of REP +1 | Start date of 'Post-study' |
| Post-study | Last date subject status obtained / last date subject known to be alive + 1 (if subject is lost to follow-up) / date of refusal + 1 day / the date subject died + 1 | During the trial: open / empty;<br>after database lock (DBL): DBL +<br>1 day |

Data recorded between the first administration of trial medication until up to 30 days (Residual effect period; REP) after the last administration of trial medication will be considered as on-treatment.

### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Even though no per protocol population is defined, subjects with potentially important protocol deviations (iPD) will be identified and documented. Potentially important protocol deviations are defined in <u>Table 6.2:1</u>. The final list of iPDs will be confirmed at the last report planning meeting (RPM) before the database lock at the time of the CTR.

If any manual iPDs are identified, they are to be summarized into categories and will be captured in the MQRM/RPM minutes via an accompanying Excel spreadsheet (3).

Table 6.2:1 Important protocol deviations

| Category/<br>Code | | Description | Comment/Example | Excluded from |
|---|---|---|---|---|
| | | | | Irom |
| A | | Inclusion/Exclusion Criteria | | |
| | A1 | Criteria related to safety | | |
| | A1.1 | Patient has condition that may cause additional risk from study medication | EX 7, EX 12, EX 19 | None |
| | A1.2 | Patient has laboratory assessments that may cause additional risk. | EX 8-11 | None |
| | A1.3 | Patient is unable to comply with the protocol | EX 13, EX 20 | None |
| | A2 | Criteria related to efficacy | | |
| | A2.1 | Patient does not have trial diagnosis or is not part of the target population | IN 1-4, EX 1, EX 2 | None |
| В | | Legal criteria | | |
| | B1 | Informed consent not available/not done | IN 5 | All |
| | B2 | Informed consent after visit 1 | IN 5 | None |
| | В3 | Men or women who are sexually active and not using adequate contraception. | EX 16, EX 17 | None |
| | B4 | Pregnant or nursing female patient | EX 15 | None |
| | B5 | Patient's age < 18 | IN 1 | None |
| C | | Administration of trial medication not in accordance with the protocol | | |
| | C1 | Administration of trial medication not in accordance with the protocol | As marked in the eCRF, review and decision at medical and quality review meetings (MQRM) / report planning meetings (RPM) | None |

Table 6.2:1 Important protocol deviations (cont.)

| Category/ | | Description | Comment/Example | Excluded |
|---|---|---|---|---|
| Code | | | | from |
| | C2 | Continuation of treatment although criteria for retreatment are not met | Create listing, decision at medical and quality review meetings (MQRM) / report planning meetings (RPM) | None |
| | СЗ | Unjustified intra-patient dose-<br>escalation | Create listing, decision at MQRM / RPM | None |
| | C4 | Withdrawal of patient not performed according to CTP | Create listing, decision at MQRM / RPM | None |
| | C5 | Discontinuation of decitabine not performed according to CTP | Create listing, decision at MQRM / RPM | None |
| | C6 | Discontinuation of BI 836858 not performed according to CTP | Create listing, decision at MQRM / RPM | None |
| D | | Restrictions | | |
| | D1 | Additional experimental anti-<br>cancer, chemo-, immuno-,<br>hormone - or radiotherapy<br>during the study or too shortly<br>before the study. | Create listing, decision at MQRM / RPM (and EX 6) | None |
| E | | Missing data | | |
| | E1 | Baseline bone marrow<br>assessment not within 14 days<br>prior to first treatment | Create listing, decision at MQRM / RPM | None |
| | E2 | Missing disease assessment at a time point where disease assessment was required | Create listing, decision at MQRM / RPM | None |

#### 6.3 SUBJECT SETS ANALYSED

Where applicable, the following subject sets will be defined for the Phase I and Phase II part separately.

- Screened set (SS): This subject set includes all subjects who have signed the informed consent. The SS will be used for subject disposition tables.
- Treated set (TS): This subject set includes all subjects who were documented to have received at least one dose of trial medication.
- MTD evaluable set: This subject set includes all subjects who were entered, treated
  and completed first cycle of planned treatment or subjects received at least 2 doses of
  BI 836858 due to BI 836858-related toxicity but not replaced.



#### 6.5 POOLING OF CENTRES

Not applicable because centre/country is not included in the statistical

### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

If not stated otherwise, missing data will not be imputed and remain missing. Potential outliers will be reported and analysed as observed.

Missing or incomplete AE dates are imputed according to BI standards (4).

For missing laboratory data at Visit 1 (before the very first administration of study medication) data from preceding visits will be used.

# 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

Study days and visits will be labelled according to the CTP's flow chart.

Unless otherwise specified, baseline is defined as the time-point closest to but prior to first administration of trial medication in course 1. Note that for some trial procedures (for example body weight, vital signs, laboratory tests) this may be the value measured on the same day trial medication was started. In these cases it will be assumed that the

measurements were taken according to protocol, i.e. prior to first intake of any trial medication.

Laboratory values: Baseline is defined as the latest time-point before the very first administration of any trial medication in course 1. For laboratories where not only the examination date but also time are recorded, examination time has to be taken into account when defining baseline. That is, a laboratory value on the same date as the first trial drug administration is considered as baseline value if and only if the time of laboratory value is before or the same as the time of first trial drug administration.

# 7. PLANNED ANALYSIS

The labelling and display format of statistical parameters will follow the guideline "Reporting of Clinical Trials and Project Summaries" (7).

For End-Of-Text (EoT) tables, the set of summary statistics is: N / Mean / Standard deviation (SD) / Min / Median / Max.

For tables that are provided for endpoints with some extreme data, median, quartiles and percentiles will be preferred to mean, standard deviation, minimum and maximum.

In general, means, medians, SD and percentiles will be presented to one more decimal place than the raw data Minima and maxima will be presented to the same number of decimal places as the raw data.

Tabulations of frequencies for categorical data will include all possible categories (even if with no count and also the missing category if there is missing data) and will display the number of observations in a category as well as the percentage (%) relative to the number of subjects in the respective treatment group (unless otherwise specified, all subjects in the respective subject set whether they have non-missing values or not). Percentages will be rounded to one decimal place. The category missing will be displayed only if there are actually missing values.

If a table presents only categorical data, "N (%)" will be displayed in the column header only.

Abbreviations (e.g., Wors.) or acronyms (e.g., PD) will not be displayed in tables and Subject Data Listings (SDLs) without any explanation. They will be either spelled out or explained in footnotes.

If applicable, conversion from days to weeks, months and years will be as follows:

- Weeks = days  $\div$  7
- Months =  $12 \times days \div 365.25$
- Years = days  $\div$  365.25

# 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Standard descriptive analyses and summary tables are planned for this section of the report. Data will be summarized by treatment group and a "total" column will be included in the summary tables.

Body Surface Area (BSA):

$$BSA[m^2] = 0.007184 \times height[cm]^{0.725} \times weight[kg]^{0.425}$$

<u>Time from first diagnosis [months]</u> = (date of informed consent - date of first diagnosis +1)[days]×12/365.25

### 7.2 CONCOMITANT DISEASES AND MEDICATION

Only descriptive statistics are planned for this section of the report.

Concomitant diseases will be coded similarly as adverse events based on the most current Medical Dictionary for Regulatory Activities (MedDRA®) version. Concomitant therapies (CTs) will be coded according to WHO DD. CTs will be classified according to the Anatomical, Therapeutic, Chemical (ATC) classification system. The third ATC level will be used to categorize CTs by therapy type. In situations where a medical product may be used for more than one equally important indication, there are often several classification alternatives. As appropriate, subjects receiving CTs with more than one possible ATC level-three category will be counted more than once; footnotes will clarify this possible double counting in tables.

### 7.3 TREATMENT COMPLIANCE

Only descriptive statistics are planned for this section of the report.

# 7.4 PRIMARY ENDPOINT(S)

#### Phase I

The primary endpoints are the MTD and the occurrence of DLT. The MTD is determined from the number of non-replaced subjects with DLT during the MTD evaluation period.

The MTD evaluation period is defined as the time from the first administration of study treatment to the start of the second treatment cycle or the end of the 30-day residual effect period after the last drug administration, whichever comes first. Subjects who were replaced during the MTD evaluation period are not considered for MTD determination. Those subjects who have completed the MTD evaluation period without having been replaced are referred to as subjects evaluable for MTD.

An overall summary of subjects with DLT(s) which occurred during the MTD evaluation period and the on-treatment period will be provided for each dose cohort.

Subjects who were treated but replaced are not considered for the MTD determination.

However, all information, including adverse events qualifying for a DLT from later times, will be considered in the final determination of the recommended Phase II dose (RP2D).

In order to describe the occurred dose escalation steps, a listing of all treated subjects will be provided. This will include the initial dose of the investigational medicinal product, subject number, treatment start date, DLT in MTD evaluation period [y/n], Evaluable for MTD [y/n] and will be sorted by treatment start date.

# 7.5 SECONDARY ENDPOINT(S)

### Phase I

The secondary endpoint overall response will be listed only. If considered useful, aggregated tables will be provided where different doses might be grouped.

#### 7.7 EXTENT OF EXPOSURE

Standard descriptive analyses over all treatment courses will be performed. This will include a summary of the variables defined in <u>Section 5.4.1</u> and will comprise a mixture of frequency and percentages, as well as summary statistics.

The time to treatment discontinuation is defined as (date of last administration of trial medication—date of randomisation + 1). Subjects who have not discontinued treatment will be censored at the earliest of the following: date of last administration of trial medication, or date of data cut-off. Subjects who are randomised, but did never receive study medication will be censored on the day of randomisation

A Kaplan-Meier plot of time to treatment discontinuation by treatment group will be presented.

### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the treated set.

# 7.8.1 Adverse Events

The analyses of adverse events (AEs) will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and NOT the number of AEs.

The analyses will be based on BI standards. Adverse events will be coded with the most recent version of MedDRA. The severity of AEs will be scaled according to CTCAE version 4.03.

Reporting will be done according to version 6 of the AE guideline (8).

TSAP for BI Trial No: 1315.2

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

For analysis of AE attributes such as duration, severity, etc. multiple AE occurrence data on the CRF, will be collapsed into AE episodes provided that all of the following applies:

- The same MedDRA lowest level term was reported for the occurrences.
- The occurrences were time-overlapping or time-adjacent (time-adjacency of 2 occurrences is given if the second occurrence started on the same day or on the day after the end of the first occurrence).
- Treatment did not change between the onset of the occurrences OR treatment changed between the onset of the occurrences, but no deterioration was observed for the later occurrence.

For each subject, all episodes with the same preferred term (PT) (system organ class, SOC) will be counted only once using a worst case approach for all AE attributes including CTCAE grading.

The analysis of adverse events will be based on the concept of treatment emergent adverse events, where a treatment emergent AE has an onset in the analysing treatment period. All adverse events occurring before first intake of trial medication will be assigned to 'screening' and all adverse events occurring after last intake of trial medication + 30 days will be assigned to 'post-treatment' (in randomized trials for listings only). For details on the treatment definition, see Section 6.1. In addition, a listing will be provided, detailing the actual treatment on the day when the adverse event started.

# Adverse events of special interest (AESIs):

Adverse events of special interest (AESIs) are defined in CTP Section 5.3.8.1 as infusion related reactions (IRRs) of CTCAE grade >= 3, DLTs (occurring during the MTD evaluation period or repeated treatment courses), tumor lysis syndrome and drug induced liver injury (DILI).

# Other significant AEs:

Other significant AEs are defined as serious and non-serious AEs that lead to dose reduction or permanent discontinuation of study medication. Their incidence will be reported by severity according to CTCAE grades.

An overall summary of adverse events will be presented. This will include the number of subjects with AEs by worst CTCAE grade. The frequency of subjects with adverse events will be summarized by treatment, primary system organ class and preferred term. The system organ classes will be sorted by default alphabetically; preferred terms will be sorted by frequency (within system organ class).

AEs leading to dose reduction, AEs leading to overall permanent discontinuation, DLTs and Adverse events of special interest (AESIs) including Infusion Related Reactions (IRRs) will be tabulated.

### Infusion related reactions (IRRs):

IRRs will be the object of special attention.

Subjects with any IRR will be tabulated by treatment and worst CTCAE grade. In addition, the number of infusions and the number of IRRs will be displayed by treatment.

The duration of IRR [h] and the time since start of the respective infusion [min] together with IRR related symptoms will be tabulated by infusion number and overall.

- Duration of IRR [h] = (End time of IRR Start time of IRR) [seconds] / 3600
- Time since start of the respective infusion [min] = (Start time of IRR Start time of infusion) [seconds] / 60

The relationship between the occurrence of IRRs and infusion rate as well as the administration of premedication will be examined.

For IRR summary, time since administration of treatment, duration of IRR, and related symptoms will be summarized descriptively by infusion timepoints.

# <u>User-defined AE categories (UDAEC)</u>

User-defined AE categories (UDAEC) are defined in in Table <u>7.8.1:1</u>. For UDAECs which contain sub-searches and/or two sensitivity levels (broad and narrow) all possibilities will be displayed on the UDAEC level in tables . For example for UDAEC "Infusion related infections" the tables will include the UDAEC "Infusion related reactions broad" and "Infusion related reactions narrow". Similarly for UDAEC "Bleeding", it will include "Bleeding - SMQ Haemorrhage", "Bleeding - SMQ Haemorrhage laboratory terms broad", "Bleeding - SMQ Haemorrhage laboratory terms narrow", "Bleeding - SMQ Haemorrhage terms (excl. laboratory terms) narrow".

Table 7.8.1:1 Definition of user-defined AE categories

| Special Search | Definition | Sensitivity |
|---|---|---|
| Category | | |
| Infusion related | SMQ 20000021 + infusion related reaction | Narrow (Algorithm) |
| reactions | PT 10051792 | |
| (hypersensitivity) | | |
| Bleeding | SMQ Haemorrhage 20000038 | Narrow & broad |
| | SMQ Haemorrhage terms (excl. laboratory terms) 20000039 | Narrow |
| | SMQ Haemorrhage laboratory terms 20000040 | Narrow & broad |
| Nausea | BIcMQ Nausea 30000078 | Narrow & broad |
| Vomiting | BIcMQ Vomiting 30000091 | Narrow & broad |

Table 7.8.1:1 Definition of user-defined AE categories (cont.)

| Special Search<br>Category | Definition | Sensitivity |
|---|---|---|
| Drug related hepatic disorders | SMQ Drug related hepatic disorders 20000006 | Narrow & broad |
| | SMQ Cholestasis and jaundice of hepatic origin 20000009 | Narrow & broad |
| | SMQ Drug related hepatic disorders - severe events only 20000007 | Narrow & broad |
| | SMQ Liver related investigations, signs and symptoms 20000008 | Narrow & broad |
| | SMQ Liver-related coagulation and bleeding disturbances 20000015 | Narrow & broad |
| ALT | BIcMQ Elevated Specific Liver Function<br>Parameters sub-search1 30000022 | Narrow & broad |
| AST | BIcMQ Elevated Specific Liver Function<br>Parameters sub-search2 30000023 | Narrow & broad |
| ALKP | BIcMQ Elevated Specific Liver Function<br>Parameters sub-search3 30000024 | Narrow & broad |
| gGT | BIcMQ Elevated Specific Liver Function<br>Parameters sub-search4 30000025 | Narrow & broad |
| Bilirubin | BIcMQ Elevated Specific Liver Function<br>Parameters sub-search5 30000026 | Narrow & broad |
| Neutropenia | BIcMQ Neutropenia 30000031 | Narrow & broad |
| Cardiac disorders <sup>1</sup> | SMQ Ischaemic heart disease 20000043 SMQ Cardiac failure 20000004 SMQ Cardiac arrhythmias 20000049 | Narrow & broad Narrow & broad Narrow & broad |
| Tumour Lysis<br>Syndrome | SMQ Tumour Lysis Syndrome 20000219 SMQ Torsade de point/QT prolongation Broad (20000001) SMQ Cardiac arrhythmia terms broad (incl bradyarrhythmias and tachyarrhythmias) (20000050) | All broad |
| Fluid accumulation | SMQ Convulsions broad (20000079) HLT Total fluid volume increased 10044085 HLT Oedema NEC 10030113 | |

Table 7.8.1:1 Definition of user-defined AE categories (cont.)

| Special Search | Definition | Sensitivity |
|---|---|---|
| Category | | |
| | HLT Pulmonary oedemas 10037424 | |
| | HLT Pneumothorax and pleural effusions | |
| | NEC 10035761 | |
| | PT Ascites 10003445 | |
| | PT Abnormal weight gain 10000188 | |
| Infections | Infections (incl. respiratory infections and | |
| | sepsis) - SOC 10021881 use label | |
| | "Infections and infestations" | |
| | Infections (incl. respiratory infections and | |
| | sepsis) - HLGT 10024970 use label | |
| | "Respiratory tract infections" | |
| | Infections (incl. respiratory infections and | |
| | sepsis) - HLT 10040054 use label "Sepsis, | |
| | bacteraemia, viraemia and fungaemia NEC" | |
| Inflamed gut | PT Enterocolitis 10014893 | |
| | PT Enterocolitis bacterial 10065206 | |
| | PT Enterocolitis fungal 10065205 | |
| | PT Enterocolitis helminthic 10065204 | |
| | PT Enterocolitis infectious 10058838 | |
| | PT Enterocolitis viral 10061841 | |
| | PT Colitis 10009887 | |
| | PT Enteritis 10014866 | |
| Acute febrile<br>neutrophilic<br>dermatosis | PT Acute febrile neutrophilic dermatosis 10000748 | |
| 1 | | |

A BIcMQ has been requested, however, as long as this is not available the terms as defined in Table <u>7.8.1:2</u> will be used.

Table 7.8.1:2 User-defined (sub-) search category of "Cardiac Failure"

| Selected PTs for Cardiac Failure |
|----------------------------------|
| Cardiac asthma |
| Cardiac failure |

Table 7.8.1:2 User-defined (sub-) search category of "Cardiac Failure" (cont.)

| Selected PTs for Cardiac Failure |
|---------------------------------------|
| Cardiac failure acute |
| Cardiac failure chronic |
| Cardiac failure congestive |
| Cardiac failure high output |
| Cardiac index decreased |
| Cardiac output decreased |
| Cardiogenic shock |
| Cardiomegaly |
| Cardiothoracic ratio increased |
| Dilatation ventricular |
| Left ventricular failure |
| Low cardiac output syndrome |
| Right ventricular failure |
| Oedema due to cardiac disease |
| Left ventricular dysfunction |
| Ejection fraction decreased |
| Cardiopulmonary failure |
| Diastolic dysfunction |
| Cardiac ventriculogram right abnormal |
| Cardiac ventriculogram abnormal |
| Cardiac ventriculogram left abnormal |
| Cardiac cirrhosis |
| Right ventricular dysfunction |
| Ventricular dysfunction |
| Cardiac resynchronisation therapy |
| Ventricular failure |
| Acute left ventricular failure |
| Acute right ventricular failure |
| Chronic left ventricular failure |
| Chronic right ventricular failure |
| Myocardial depression |
| Ventricular dyssynchrony |
| Systolic dysfunction |
| Neonatal cardiac failure |

UDAEC will by summarized by dose cohort, search categories and preferred terms, and CTCAE grade. Some events contribute to more than one UDAEC. Patients with such AEs are counted in each of the UDAEC but are counted only once in the overall number of patients with an AE in any UDAEC.

# Tumor Lysis Syndrome

In patients with a high tumor burden who are exposed to a highly effective therapy, there is a risk of rapid tumor destruction resulting in Tumor Lysis Syndrome (TLS).

Patients will be identified as having potential Tumor Lysis Syndrome if they met **both** of the following two criteria:

- (1) Two or more of the laboratory parameters meet the criteria in <u>Table 7.8.1:3</u>,
  - a. time window
    - i. on the day of BI 836858 infusion or the following 6 days,
    - ii. at least two of the qualifying lab values must have occurred with the same 24 hour period
- (2) Have an adverse event identified by the any of the SMQ in <u>Table 7.8.1:4</u> or have a qualifying creatinine value
  - a. Time windows: AE onset or creatinine observation at any time during the treatment or residual effect periods

Table 7.8.1:3 Laboratory Signs of Cell Destruction

| Laboratory parameter | Abnormal value |
|---|---|
| Uric acid | ≥476 µmol/L AND increase from relative baseline <sup>1</sup> by ≥25% |
| Potassium | value ≥ 6.0 mmol/L AND relative baseline < 6.0 mmol/L |
| Inorganic phosphate | ≥1.45 mmol/L AND increase from relative baseline by ≥25% |
| Calcium | <7 mg/dL² AND decrease from relative baseline by ≥25% |

<sup>&</sup>lt;sup>1</sup>Relative baseline is derived separately for each BI 836858 infusion as the last value prior to that BI 836858 infusion. Relative baseline will be derived independently for the four parameters, ie. four baseline values do not necessarily have to be derived from the same laboratory assessment.

Table 7.8.1:4 Clinical Signs of Cell Destruction

| Criterion |
|--------------------------|
| TLS broad SMQ [20000219] |

<sup>&</sup>lt;sup>2</sup>For calcium, 0.25\* mg/dL= mmol/L

Table 7.8.1:4 Clinical Signs of Cell Destruction (cont.)

### Criterion

Torsade de point/QT prolongation broad SMQ [20000001]

Cardiac arrhythmia terms broad SMQ (incl bradyarrhythmias and tachyarrhythmias) [20000050]

Convulsions broad SMQ [20000079]

Creatinine

Absolute increase from relative baseline by 26.5  $\mu$ mol/L AND increase from relative baseline by  $\geq$ 50%

For AEs during the post-treatment period, only subjects with drug related serious adverse event and protocol-specified AEs of special interest by treatment will be presented in listing.

# 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards (9). It will include a graphical summary highlighting potential cases of Hy's Law.

The analysis of laboratory data will use the same 'analysing treatments' as described for the AEs, except for that the baseline laboratory value will be included in the 'on-treatment period'. Subjects having at least one post-baseline laboratory value will be displayed in the descriptive analyses. The following parameters are of particular interest:

- haematology: haemoglobin, white blood cell count, Absolute Neutrophil Counts, platelets
- Biochemistry: aspartate transferase, alanine transferase, bilirubin, serum creatinine, urea, sodium, potassium, magnesium
- Coagulation: international normalised ratio, partial thromboplastin time

<u>Laboratory values</u>: Baseline is defined as the latest time-point before the very first administration of study medication. A laboratory value on the same date as the first study drug administration is considered as according to protocol, i.e. as prior to first study drug administration and will therefore be used as baseline value.

The following outputs will be presented:

TSAP for BI Trial No: 1315.2

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Worst CTCAE grade experienced during the on-treatment phase.
- Transitions of CTCAE grade from baseline to worst laboratory value, from worst to last laboratory value on treatment and from baseline to last laboratory value during the on-treatment phase.

Worst laboratory value and its CTCAE grade (highest CTCAE grade) over all courses will be calculated for each laboratory parameter specified above.

The last laboratory value on treatment is the laboratory value of the last visit of the last course of each subject.

Furthermore, a summary table of possible clinically significant abnormalities will be given.

Possible clinically significant abnormal laboratory values are defined as those laboratory values that are of CTCAE grade  $\geq 2$  and show an increase from baseline value by at least one CTCAE grade. Frequency of subjects with possible clinically significant abnormal laboratory values will be provided whenever applicable. If no baseline value is available but the subject has a post-baseline laboratory value of CTCAE grade  $\geq 2$  an increase from baseline will be assumed, i.e. the laboratory value considered as possible clinically significant.

## Hepatic injury:

As defined in the CTP a hepatic injury (DILI) is defined by the following alterations of hepatic laboratory parameters:

- an elevation of AST and/or ALT >3 fold ULN combined with an elevation of total bilirubin >2 fold ULN measured in the same blood draw sample, and/or
- marked peak aminotransferase (ALT, and/or AST) elevations ≥10 fold ULN

Potential Hepatic enzyme elevations (potential Hy's law cases): These are defined as those cases where a combination of all of the following events occurred: any on-treatment value of ALT and/or AST > 3ULN with total bilirubin ≥ 2ULN and ALKP < 2ULN. The events can occur in any order, but must occur within 14 days of the previous event, i.e. the second event must occur within 14 days of the first event, and the third event must occur within 14 days of the second event, etc. Subjects with missing laboratory values for liver enzymes will be excluded from these analyses.

In addition, eDISH plot will be by plotted to display the maximum on-treatment AST/ALT and maximum bilirubin in terms of ULN.

Neutrophil and platelet counts of each patients will be plotted in log scale graphs.

# 7.8.3 Vital signs

Only descriptive statistics are planned for vital sign report. Observed value and change from baseline values will be summarized.

#### 7.8.4 **ECG**

12-lead resting ECGs are done throughout the study and are assessed for pathological results which are to be recorded as either concomitant disease or AE by the Investigator. ECG results will be listed.



#### 8. **REFERENCES**

| 1 | CPMP/ICH/363/96: "Statistical Principal for Clinical Trials", ICH Guideline Topic E9 Step 5; Note For Guidance on Statistical Principal for Clinical Trials, current version, EMA webpage. |
|---|---|
| 2 | 001-MCS-50-415_RD-01: "TSAP annotations", current version; IDEA for CON. |
| 3 | 001-MCS-40-413: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON. |
| 4 | BI-KMED-BDS-HTG-0035: "Handling of missing and incomplete AE dates", current version; KMED. |
| 5 | 001-MCS-36-472: "Standards and processes for analyses performed within Clinical Pharmacokinetics/Pharmacodynamics", current version; IDEA for CON. |
| 6 | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON. |
| 7 | 001-MCS-50-415: "Clinical Trial Data Analysis", current version; IDEA for CON. |
| 8 | <i>BI-KMED-BDS-HTG-410</i> : "Analysis and Presentation of Adverse Event Data from Clinical Trials", KMED. |
| 9 | <i>BI-KMED-BDS-HTG-0042</i> : "Handling, Display and Analysis of Laboratory Data", current version; KMED . |



#### **HISTORY TABLE 10.**

History table Table 10: 1

| Version | Date<br>(DD-MMM-<br>YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Initial | 14-Jul-16 | | None | This is the initial TSAP with necessary information for trial conduct. |
| Final | 19-Nov-19 | | None | This is the final TSAP. |